CLINICAL TRIAL: NCT02653183
Title: A Prospective, Randomized, Controlled Clinical Investigation, Comparing Two Postoperative Wound Dressings Used After Elective Hip and Knee Replacement
Brief Title: Prospective, Randomized Clinical Investigation of Two Different Postoperative Wound Dressings
Acronym: MxBPo02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MxB Po 02
Record Dates: First submitted 2015-12-11; First posted 2016-01-12 (Estimated); Results first posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2017-09

CONDITIONS: Hip Surgery Corrective; Knee Injuries
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Device Aquacel Surgical (Active Comparator): Aquacel Surgical is a sterile, one piece post-operative dressing from Convatec.
  Duration of treatment:
  Total 5 days included the day of surgery and 4 post-operative days.
  Interventions: Device: Experimental: Mepilex Border Post-Op
- Device Mepilex Border Post-Op (Experimental): Post-operative all-in-one self-adherent soft silicone coated foam dressing.
  Duration of treatment:
  Total 5 days included the day of surgery and 4 post-operative days.
  Interventions: Device: Active Comparator: Aquacel Surgical

INTERVENTIONS:
Device: Active Comparator: Aquacel Surgical — Post-operative all-in-one self-adherent soft silicone coated foam dressing. Duration of treatment: Total 5 days included the day of surgery and 4 post-operative days.
  Arms: Device Mepilex Border Post-Op
Device: Experimental: Mepilex Border Post-Op — Aquacel Surgical is a sterile, one piece post-operative dressing.Duration of treatment:
  Total 5 days included the day of surgery and 4 post-operative days.
  Arms: Device Aquacel Surgical

SUMMARY:
The primary objective of this investigation is to evaluate if complications related to surgical wound are more common in the treatment group compared to the control group starting from operation day until last visit.

The secondary objectives are to evaluate:

* the performance of the dressing
* the comfort, conformability and the acceptability of the dressing
* pain before and during dressing removal on the last visit

DETAILED DESCRIPTION:
A prospective, randomized clinical investigation will be conducted at two to three sites in Belgium and Sweden.

Male or female, 18 years and older undergoing primary hip or knee arthroplasty with an expected hospital stay of 4 days or longer will be included in to the clinical investigation.

100 evaluable patients (i.e. 50 subjects per arm). The treatment arm (either Mepilex Border Post-Op or Aquacel Surgical) Patient eligibility will be established before treatment randomization. Patients will be randomized using optimal allocation (minimization) balancing for the following baseline variables type of surgery (hip or knee), age and skin status. Eligible patients will be randomized to receive Mepilex Border Post-Op or Aquacel surgical in a ratio of 1:1 provided.

ELIGIBILITY:
Inclusion Criteria, enrolment phase

1. Age ≥ 18 years
2. Have an expected total length of stay of 4 postoperative days or more
3. Plan for elective primary arthroplasty of the hip or knee
4. Plan for incision size > 18 cm
5. Give their written informed consent to participate

Inclusion Criteria, randomization phase

1. Undergoing elective primary arthroplasty of the hip or knee

Exclusion Criteria,enrolment phase

1. Known allergy or hypersensitivity to any of the components of the dressings
2. Multitrauma
3. Undergoing arthroplasty due to tumour
4. Wound at the surgical site prior to surgery
5. Neurological deficit of operated side ,hemiplegia, etc.
6. Documented skin disease at time of enrolment, as judged by the investigator
7. Previously enrolled in the present investigation
8. Included in another ongoing investigation at present which can interfere with the result of the dressing, judged by the investigator
9. Involvement in the planning and conduct of the clinical investigation, applies to all Molnlycke Health Care staff, investigational site staff and third party vendor.

Exclusion Criteria, randomization phase

1. Dressing size does not fit the incision area, over 18 cm
2. Complications that would increase wound risks if investigation dressing is applied
3. Postoperative drain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (2):
  - University Hospital Gent, Belgium, Ghent
  - Medisch Centrum Latem, Sint-Martens-Latem
- Södersjukhuset, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 118 subjects were enrolled and 113 subjects were randomized, Out of the 113 randomized subjects. Screening failure, IP never applied, inclusion criteria inclusion criteria 4 not met.=5 Not included in the analysis The patient signed IC after data been entered into the eCRF. Excluded from the analysis=5
Groups:
- Device Mepilex Border Post-Op: Post-operative all-in-one self-adherent soft silicone coated foam dressing.
  Active Comparator: Aquacel Surgical: Post-operative all-in-one self-adherent soft silicone coated foam dressing
- Device Aquacel Surgical: Aquacel Surgical is a sterile, one piece post-operative dressing from ConvaTec.
  Experimental: Mepilex Border Post-Op: Aquacel Surgical is a sterile, one piece post-operative dressing
Period: Overall Study
Arm/Group | Device Mepilex Border Post-Op | Device Aquacel Surgical
Started | 53 | 50
Completed | 49 | 46
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Device Mepilex Border Post-Op | Device Aquacel Surgical | Total
Number analyzed (Participants) | 53 | 50 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 16 | 31
  >=65 years | 38 | 34 | 72
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 27 | 63
  Male | 17 | 23 | 40
Type of surgery [Number; unit: participants]
  Hip | 26 | 25 | 51
  Knee | 27 | 25 | 52
Skin type [Number; unit: participants]
  Normal | 45 | 41 | 86
  Dry | 5 | 4 | 9
  Oily | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Composite Variable Ranging From 0 to 7, Combining Complications (Dressing Failure) Related Surgical Wound, Computed as: 3*(Dressing Change) + 2*Blister + (Pain>=30mm) + Redness on the Skin Under the Dressing
Description: Scale range from 0 (no dressing failure) to 7 ( complete dressing failure).
Time Frame: 0-5 days
Measure: Number; unit: participants
Arm/Group | Device Mepilex Border Post-Op | Device Aquacel Surgical
Number analyzed (Participants) | 53 | 50
participants
  Composite score 0 | 36 | 32
  Composite score1 | 10 | 11
  Composite score 2 | 0 | 1
  Composite score 3 | 4 | 4
  Composite score 4 | 3 | 1
  Composite score 5 | 0 | 1

2. Secondary Outcome: Dressings Adherence to the Staples/Sutures
Description: Dressings adherence to the staples/sutures? Yes/No
Time Frame: 0-5 days
Measure: Number; unit: participants
Arm/Group | Device Mepilex Border Post-Op | Device Aquacel Surgical
Number analyzed (Participants) | 53 | 50
participants
  No | 53 | 50
  Yes | 0 | 0

3. Secondary Outcome: Itching Feeling Under the Dressing
Description: Itching feeling under the dressing? Yes/No
Time Frame: 0-5 days
Measure: Number; unit: participants
Arm/Group | Device Mepilex Border Post-Op | Device Aquacel Surgical
Number analyzed (Participants) | 53 | 50
participants
  No | 53 | 48
  Yes | 0 | 2

4. Secondary Outcome: Patients Satisfaction With Wearing the Dressing
Description: 4 point rating scale ( poor, good, very good,excellent)
Time Frame: 0-5 days
Measure: Number; unit: participants
Arm/Group | Device Mepilex Border Post-Op | Device Aquacel Surgical
Number analyzed (Participants) | 53 | 50
participants
  Poor | 0 | 1
  Good | 13 | 19
  Very good | 22 | 24
  Excellent | 18 | 6

5. Secondary Outcome: Nurses/Doctors Satisfaction With Applying the Dressing
Description: 4 point rating scale ( poor, good, very good,excellent)
Time Frame: 0-5 days
Measure: Number; unit: participants
Arm/Group | Device Mepilex Border Post-Op | Device Aquacel Surgical
Number analyzed (Participants) | 53 | 50
participants
  Poor | 2 | 2
  Good | 13 | 35
  Very Good | 17 | 12
  Excellent | 21 | 1

6. Secondary Outcome: Patients Mobility After Operation
Description: 4 point rating scale ( poor, good, very good,excellent)
Time Frame: 0-5 days
Measure: Number; unit: participants
Arm/Group | Device Mepilex Border Post-Op | Device Aquacel Surgical
Number analyzed (Participants) | 53 | 50
participants
  Poor | 0 | 1
  Good | 12 | 19
  Very good | 23 | 24
  Excellent | 18 | 6

7. Secondary Outcome: Local/Systemic Infection
Description: Local/systemic infection? Yes/No
Time Frame: 0-5 days
Measure: Number; unit: participants
Arm/Group | Device Mepilex Border Post-Op | Device Aquacel Surgical
Number analyzed (Participants) | 53 | 50
participants
  No | 53 | 50
  Yes | 0 | 0

8. Secondary Outcome: Pain Level Before and During Dressing Removal
Description: Different adhesive on the dressings, can any difference be identified during dressing removal.
  Pain level before dressing removal and pain level during dressing removal. Only measured on the last visit, with this point, the patient has not so much pain from the hip/knee joint replacement, which can have an effect on the result of dressing removal pain VAS scale (0-100 mm) 0= No pain, 100= Moste intense pain imainable.
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Device Mepilex Border Post-Op | Device Aquacel Surgical
Number analyzed (Participants) | 53 | 50
units on a scale
  Pain before removal of dressing at last visit | 7.8 (13.8) | 4.9 (6.3)
  Pain during removal of dressing at last visit | 6.9 (11.7) | 10 (12)

ADVERSE EVENTS:
Arm/Group | Device Mepilex Border Post-Op | Device Aquacel Surgical
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/50
Other Adverse Events (participants affected / at risk) | 22/53 | 15/50
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Device Mepilex Border Post-Op (N=53) | Device Aquacel Surgical (N=50)
Nausea (Surgical and medical procedures) | 9 | 8
Obstipation (Surgical and medical procedures) | 5 | 1
Allergic reaction (Surgical and medical procedures) | 0 | 1
Dizziness (Surgical and medical procedures) | 1 | 0
Elevated glucose levels (Surgical and medical procedures) | 2 | 2
Excema, medication related (Surgical and medical procedures) | 1 | 0
Fever (Surgical and medical procedures) | 1 | 1
Insomnia (Surgical and medical procedures) | 0 | 1
Itching (Surgical and medical procedures) | 0 | 1
Low hemoglobine level (Surgical and medical procedures) | 1 | 0
Skin allergy (Surgical and medical procedures) | 1 | 0
Confusion (Surgical and medical procedures) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other